CLINICAL TRIAL: NCT00664014
Title: Randomized, Double-blind, Multicenter, Placebo-controlled (Standard Therapy + Placebo), Phase 2 Efficacy and Safety Study of the Tolvaptan Tablets in Patients With Non-hypovolemic Non-acute Hyponatremia
Brief Title: A Phase 2 Efficacy and Safety Study of the Tolvaptan Tablets in Patients With Non-hypovolemic Non-acute Hyponatremia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Beijing Research Institute (Industry)
Collaborators: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 156-07-802-01
Record Dates: First submitted 2008-04-14; First posted 2008-04-22 (Estimated); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Hypovolemic Hyponatremia
Keywords: hyponatremia; Non-acute and non hypovolemic hyponatremia
MeSH Terms: conditions — Hyponatremia | interventions — Tolvaptan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tolvaptan (Experimental)
  Interventions: Drug: Tolvaptan
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tolvaptan — Tablet;15mg/tab;15/30/60mg/day for 7days Plus conventional therapy according to each patient's underlying disease, such as congestive heart failure, hepatic cirrhosis and SIADH or others.
  Arms: Tolvaptan
Drug: Placebo — placebo plus conventional therapy according to each patient's underlying disease, such as congestive heart failure, hepatic cirrhosis and SIADH or others.
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, multicenter, placebo-controlled (standard therapy + placebo), phase 2 efficacy and safety study of the Tolvaptan tablets in treatment of patients with non-hypovolemic non-acute hyponatremia arising from a variety of etiologies. 240 (120 in each group) patients are to be enrolled randomly into Tolvaptan group or placebo group. Subjects in Tolvaptan group will receive standard therapy + Tolvaptan (15-60mg/day), while those in control group receiving standard therapy + placebo. The starting dose of tolvaptan is 15mg and it could be titrated up to 30mg and then,if necessary, to the maximum of 60mg according to a certain titration scheme based on patients' response of serum sodium level. The study includes a 2-day screening period from day -2 to day -1, 7-day inpatient study treatment (day 1 to day 7 ). After study treatment, subjects will be Followed-up on safety events on day 14 - 16. The Primary Efficacy Variable is the change of serum sodium from baseline. For patients with Congestive Heart Failure (CHF) or hepatic cirrhosis, change of body weight, fluid balance and symptoms improvement of CHF and hepatic edema will be assessed as secondary efficacy variables.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent.
2. Age:18～75 (when informed consent is obtained)，male or female.
3. Non-hypovolemic and non acute hyponatremia with a Serum sodium < 135mEq/L before randomization. (main underlying diseases include CHF, hepatic cirrhosis with edema, SIADH and others)
4. In-patient subjects.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2008-05; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
The change of average daily Area Under the Curve (AUC) of serum sodium by day 4 and 7 comparing with baseline serum sodium level within the double-blind therapy period. | 4 and 7 days

SECONDARY OUTCOMES:
For CHF and hepatic edema patients, improvement of symptoms and relevant physical examination measures or ultrasound test findings . Other secondary efficacy variables on blood serum sodium, fluid balance or body weight change. | 4 or 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Wenling Zhu, Principal Investigator — Peking Union Medical College Hospital; Feng Gu, Principal Investigator — Peking Union Medical College Hospital; Jidong Jia, Principal Investigator — Beijing Friendship Hospital
Locations (13):
- China (13):
  - Department of Cardiology, the Third Xiangya Hospital, Central South University, Changsha, Hunan
  - Department of Cardiology, Xiangya Hospital, Central South University, Changsha, Hunan
  - Cardiology, Jilin University Second Hospital, Changchun, Jilin
  - Endocrinology, West China Hospital Sichuan University, Chengdu, Sichuan
  - Cardiology / Endocrinology, Peking Union Medical College Hospital, Beijing
  - Cardiology / Hepatology, Beijing Friendship Hospital, Beijing
  - Cardiology/Endocrinology/Infection, Beijing University First Hospital, Beijing
  - Endocrinology, No. 301 hospital, Beijing
  - Hepatology, Beijing Renmin Hospital, Beijing
  - Hepatology/Endocrinology, Chongqing Medical University Second Hospital, Chongqing
  - Hepatology / Endocrinology, Shanghai Changzheng Hospital, Shanghai
  - Cardiology, Tianjin Medical University Second Hospital, Tianjin
  - Endocrinology, Tianjin General Hospital, Tianjin

REFERENCES:
- [Derived] Wang S, Zhang X, Han T, Xie W, Li Y, Ma H, Liebe R, Weng H, Ding HG. Tolvaptan treatment improves survival of cirrhotic patients with ascites and hyponatremia. BMC Gastroenterol. 2018 Sep 4;18(1):137. doi: 10.1186/s12876-018-0857-0. PMID 30180806
- [Derived] Chen S, Zhao JJ, Tong NW, Guo XH, Qiu MC, Yang GY, Liu ZM, Ma JH, Zhang ZW, Gu F. Randomized, double blinded, placebo-controlled trial to evaluate the efficacy and safety of tolvaptan in Chinese patients with hyponatremia caused by SIADH. J Clin Pharmacol. 2014 Dec;54(12):1362-7. doi: 10.1002/jcph.342. PMID 24906029